CLINICAL TRIAL: NCT02306486
Title: The Effect of Oxalic Acid on Cervical Restorations on Hypersensitive Teeth, a Double-blind Randomized Controlled Clinical Trial. One Year Follow up
Brief Title: The Effect of Oxalic Acid on Cervical Restorations
Acronym: OxalicAc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Prof.Eduardo Fernández G., University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/03
Record Dates: First submitted 2014-11-24; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- z250 resin composite (Placebo Comparator): (n=31) Treated with distilled water (placebo) and restored with a methacrylate resin-based-composite (Z250, 3M ESPE, shade: A3)
- z250 resin composite + oxalic acid (Active Comparator): (n=31) treated with 0.5% oxalic acid (Desenssiv, SSWhite)(intervention)// and restored with a methacrylate resin-based-composite (Z250, 3M ESPE, shade: A3)
  Interventions: Other: with 0,5% oxalic acid (Desenssiv SSWhite)
- p 90 resin composite (Placebo Comparator): (n=31) Treated with distilled water (placebo) and restored with a silorane resin-based-composite.
- p 90 resin composite + oxalic acid (Active Comparator): (n=31) treated with 0,5% oxalic acid (Desenssiv SSWhite)(Intervention)/ and restored with a silorane resin-based-composite (Filtek Silorane p90, £M ESPE, shade:)
  Interventions: Other: with 0,5% oxalic acid (Desenssiv SSWhite)

INTERVENTIONS:
Other: with 0,5% oxalic acid (Desenssiv SSWhite) — with 0,5% oxalic acid (Desenssiv SSWhite) , desensitizer for sensivity cervical lesions on tooth
  Other Names: Desenssiv SSWhite
  Arms: p 90 resin composite + oxalic acid; z250 resin composite + oxalic acid

SUMMARY:
The aim of this double-blind randomized controlled clinical trial was to evaluate the effect on dentin sensitivity using oxalic acid desensitizing agent before restoring with resin-based-composites, during one-year follow-up. One hundred and twenty two cervical lesions (31 patients, age range between 24 and 66 years) were selected and randomly divided into four groups: OA/Z250: treated with acid oxalic desensitizing agent (Desenssiv, SSWhite) before restoring with a methacrylate resin-based-composite (Z250, 3M ESPE), (n=31), OA/P90 treated with acid oxalic desensitizing agent (Desenssiv, SSWhite) before restoring with a silorane resin-based-composite (Silorane p90, 3M ESPE) (n=31), Z250 restored with methacrylate resin-based-composite (Z250, 3M ESPE) (n=30) and P90 restored with a silorane resin-based-composite (Silorane p90, 3M ESPE) (n=30). All lesions were evaluated at baseline, immediately and 1, 2, 3, 6 months and 1 year after treatment. Teeth sensitivity was measured by visual analog scale (VAS) after evaporation and tactile stimuli

DETAILED DESCRIPTION:
The study design was a split-mouth placebo-controlled randomized clinical trial according to CONSORT recommendations. Patients were recruited in the Clinic of Dental School of University of Chile according to inclusion criteria.All patients signed the informed consent approved by the Ethics Committee (Dental School, Universidad de Chile).

Inclusion criteria were:

* Patients older than 18 years old having at least 4 teeth with cervical buccal lesions sensitive to tactile and thermal/evaporation stimuli. (moderate / severe pain by EVA)
* Teeth with surface loss on the buccal cervical area with indication of resin-composite-based restoration.

Exclusion criteria were:

* Systemic diseases related to chronic pain
* Pregnancy
* Recent periodontal surgery, orthodontic treatment or desensitizing treatment within the last 3 months.
* In treatment with NSAIDs
* Teeth with caries or restorations
* Incisor teeth (to avoid cross innervation).

At baseline, two calibrated examiners (kappa >0,75) evaluated teeth sensitivity. Tactile stimulus consisted of probing the buccal cervical surface of the teeth with North-Carolina periodontal probe (Hu-Friedy). Evaporation stimulus consisted in direct air pressure application with three-in-one syringe for one second at 60 psi at room temperature, perpendicular to the tooth, 1 cm away from the surface, protecting the adjacent teeth with cotton rolls. Patients quantified their pain caused by both stimuli through VAS (Visual Analogue Scale).

Pocock method was used to allocate the groups, so they presented similar distribution according to VAS (visual analogue scale) results recorded at baseline.

The assigned groups were:

* Z250 (n=30) Treated with distilled water (placebo) and restored with a methacrylate resin-based-composite (Z250, 3M ESPE, shade: A3)
* P90 (n=30) Treated with distilled water (placebo) and restored with a silorane resin-based-composite.
* OA/Z250 (n=31) treated with 0.5% oxalic acid (Desenssiv, SSWhite) and restored with a methacrylate resin-based-composite (Z250, 3M ESPE, shade: A3)
* OA/P90 (n=31) treated with 0,5% oxalic acid (Desenssiv SSWhite) and restored with a silorane resin-based-composite (Filtek Silorane p90, £M ESPE, shade:) Blinding Oxalic acid and distilled water were applied with micro brush, brushing for 1 minute, and then rinsed with water. Restorations were made following manufacturer instructions. The adhesive system Single Bond 2 (3M ESPE) was used with resin-based-composite Z250 and its own adhesive system was used for Filtek Silorane P90. To ensure the double-blind aspect of the trial, bottles of oxalic acid and distilled water were covered so operator could not recognized them, and the same was done with both types of resin-based-composites. Patients were also not aware of which tooth corresponded with which treatment.

Clinical evaluations The same two clinical examiners, than at baseline, evaluated teeth sensitivity after 30, 60, 90, 180 and 360 days of placing the restorations. Response of pain scored with VAS was recorded after tactile and evaporation stimuli. This was performed in the same manner than at baseline, but the tactile stimulus was performed probing around the tooth/restoration margin with North-Caroline periodontal probe (Hu-Friedy).

Statistical analysis The sample size was calculated with a statistical power (0.95) considering the sensitivity by EVA as principal outcome, with a confidence level (95%) resulting in n=28 , considering the reported drop-out was added a 5%.

SPSS (SPSS, Chicago, IL, USA) was used for the statistical analyzes of this study. Differences between groups were analyzed with Wilcoxon and Mann-Whitney test. For the multiple comparisons between groups was used Friedman test. The significance level of this study was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old having at least 4 teeth with cervical buccal lesions sensitive to tactile and thermal/evaporation stimuli. (moderate / severe pain by EVA)
* Teeth with surface loss on the buccal cervical area with indication of resin-composite-based restoration.

Exclusion Criteria:

--Systemic diseases related to chronic pain

* Pregnancy
* Recent periodontal surgery, orthodontic treatment or desensitizing treatment within the last 3 months.
* In treatment with NSAIDs
* Teeth with caries or restorations
* Incisor teeth (to avoid cross innervation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
teeth sensitivity by EVA | 30 days
  days after of placing the restorations
teeth sensitivity by EVA | 60 days
  days after of placing the restorations
teeth sensitivity by EVA | 90 days
  days after of placing the restorations
teeth sensitivity by EVA | 180 days
  days after of placing the restorations
teeth sensitivity by EVA | 360 days
  days after of placing the restorations

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Fernandez, Prof., Principal Investigator — University of Chile

REFERENCES:
- [Background] Barrientos C, Xaus G, Leighton C, Martin J, Gordan VV, Moncada G. Oxalic acid under adhesive restorations as a means to reduce dentin sensitivity: a four-month clinical trial. Oper Dent. 2011 Mar-Apr;36(2):126-32. doi: 10.2341/09-364-C. PMID 21777095